CLINICAL TRIAL: NCT05400525
Title: University of Roehampton
Brief Title: Supplementation of YMETA, on Gut Health, Immunity and Metabolism in Pre-diabetic Adult Population
Acronym: YMETA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roehampton (Other)
Collaborators: Vemico Ltd. (Industry)
Responsible Party: Principal Investigator, DR ADELE COSTABILE, READER IN NUTRITION, University of Roehampton
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: LSC 22/374
Record Dates: First submitted 2022-05-27; First posted 2022-06-01 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Pre-diabetes
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- YMETA (Active Comparator): Y META is a combination of gut health focused bioactives that target both the metabolic activity of existing microbiota (Bifidobacterium spp. targeting prebiotic galacto-oligosaccharides mixture)
  Interventions: Dietary Supplement: YMETA
- Maltodextrin (Placebo Comparator)
  Interventions: Other: Placebo control

INTERVENTIONS:
Dietary Supplement: YMETA — 1 sachet containg a total of 3g i.e. 2.5g Galacto-oligosaccharides, 0.5g Bifidobacterium polysaccharides (daily)
  Arms: YMETA
Other: Placebo control — 3g Maltodextrin (i.e. DE 10) daily
  Arms: Maltodextrin

SUMMARY:
Type 2 diabetes mellitus (T2DM) is a major non-communicable disease and one of the world's fastest growing health problems. According to a 2019 report, about 463 million adults worldwide currently have diabetes and future projections indicate the number of diabetic patients will reach 700 million by 2045.1 T2DM is associated with significant morbidity, including increased risk of cardiovascular diseases (CVD) and stroke, hypertension, retinopathy and blindness, renal failure, and leg amputation. These place an enormous burden on individuals, society and the healthcare system.2

T2DM is a non-reversible but preventable condition with overweight and obesity being major risk factors. The onset of T2DM is gradual, with most individuals progressing from normoglycaemia through a pre-diabetic state. People with pre-diabetes, defined as having impaired fasting glucose (IFG), impaired glucose tolerance (IGT) or impaired glycated haemoglobin (HbA1c),2 are at increased risk of developing T2DM and its associated complications, such as CVD and retinopathy, which can develop even in the absence of progression to overt T2DM.3-5 Pre-diabetes is a prevalent and potentially reversible condition that provides an important window of opportunity for healthcare providers to implement interventions that can delay or prevent T2DM and its complications.

A substantial body of literature has provided evidence for the role of gut microbiota in metabolic diseases including type 2 diabetes.6 Indeed, there is evidence for the effects of microbiota on glucose metabolism in both preclinical animal models of T2D and in healthy animals, by means of increasing the number of inflammatory mediators, chronic inflammation, insulin resistance and increased energy intake. Among the commonly reported findings, Bifidobacterium spp appears to be the most consistently supported by the literature genus containing microbes potentially protective against T2DM. Indeed, nearly all papers report a negative association between this genus and T2DM;7-14 while only one paper reported opposite results.15

In view of the correlation between gut microbiota, more specifically Bifidobacterium spp., and diabetes, the Bifidobacterium population and their metabolic action can be taken as an important target for interventions to prevent and/or delay the development of T2DM.

DETAILED DESCRIPTION:
Y META is a combination of gut health focused bioactives that target both the metabolic activity of existing microbiota (Bifidobacterium spp. targeting prebiotic galacto-oligosaccharides mixture) and the crosstalk of existing microbiota with host mucosal immune system through gut microbiota derived signalling molecules (Bifidobacterium derived polysaccharides commercially available as Y SKIN) that interact with the gut mucosal immune system to promote its regulatory activity and prevent accumulation of gut derived chronic inflammation, in order to revert insulin resistance, the main risk factor for the development of T2DM, without the need to modify the microbiota composition with live bacteria.

In this study, we aim to explore whether a gut health focused intervention, in the form of Y META, affect blood glucose level and risk factors for diabetes in pre-diabetic subjects via modification of insulin sensitivity and other post-interventional effects.

ELIGIBILITY:
Inclusion criteria

* Adults aged between 18 and 60 years, with
* Fasting blood glucose level of 5.6-6.9mmol/L or
* Impaired HbA1c (HbA1c level of 5.7%-6.4%)
* For intervention purposes, eligible participants are also required to have a mobile phone and be able to read and speak English.

Exclusion criteria

* People with a current diagnosis or clinical history of T2DM
* People with comorbid conditions that may limit participation in the study, such as a history of an acute cardiovascular event, uncontrolled hypertension, cancer or major psychiatric or cognitive problems
* People who are already participating in a weight loss programme
* People receiving drug treatment for pre-diabetes (eg, metformin)
* People with a history of long-term use of medicines known to influence glucose metabolism (eg, corticosteroids)
* People with elevated liver enzymes (alanine aminotransferase ≥300 IU/L, aspartate aminotransferase ≥300 IU/L)
* People who take antibiotics or bacterial agents (Probiotics) within 1 month
* Pregnant women, women ready for pregnancy, and nursing mothers

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-06-10 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
Changes in blood glucose levels | Changes from baseline to 6 and 12 weeks of the intervention
  To investigate the effects of Y Meta intervention on blood glucose levels of pre-diabetics
Changes in insulin sensitivity | Changes from baseline to 6 and 12 weeks of the intervention
  To investigate the mediating effect of Y META on insulin sensitivity in pre-diabetics
Changes in gut microbiota composition | Changes from baseline to 6 and 12 weeks of the intervention
  To investigate the effect of Y META intervention on gut microbiota composition
Changes in immune response | Changes from baseline to 6 and 12 weeks of the intervention
  To investigate the effect of Y META intervention on immune function in pre-diabetics

SECONDARY OUTCOMES:
Dietary Habits | Changes from baseline to 6 and 12 weeks of the intervention
  To investigate the effect of Y META intervention on dietary habits

CONTACTS AND LOCATIONS:
Overall Officials: ADELE COSTABILE, DR, Study Director — University of Roehampton
Locations (1):
- Health Sciences Research Centre, Life Sciences Department, University of Roehampton, London, UK, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Study Protocol — https://discoverthesecretofgoodhealth.weebly.com